CLINICAL TRIAL: NCT03119441
Title: The Efficacy of Dental Water Jet in Plaque Removal During Orthodontic Treatment With Fixed Appliances: A Randomized Controlled Trial
Brief Title: Effect of Dental Waterjet on Oral Hygiene for Patients With Braces
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Responsible Party: Principal Investigator, Omar Alkadhi, Assistant professor, Riyadh Colleges of Dentistry and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FRP/2016/115
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Oral Hygiene
MeSH Terms: interventions — Dental Devices, Home Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dental water jet (Experimental): Dental water jet (Jetpik JP210)
  Interventions: Device: Dental Water Jet
- Dental floss (Active Comparator): Dental floss
  Interventions: Device: Dental Floss

INTERVENTIONS:
Device: Dental Water Jet — Dental Water Jet will be used by subjects to clean their teeth in the interproximal areas.
  Arms: Dental water jet
Device: Dental Floss — Dental Floss will be used by subjects to clean their teeth in the interproximal areas.
  Arms: Dental floss

SUMMARY:
The aim of this study is to assess the efficacy of dental water jet in plaque removal and gingival health during orthodontic treatment with fixed appliances.

DETAILED DESCRIPTION:
Subjects will be randomized into two groups. The first group will receive a dental water jet and the second group will receive dental floss. Plaque accumulation using plaque index and gingival health using gingival index will be measured at baseline and after four weeks for each group and then, results will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Subjects having orthodontic fixed appliance.
* Subjects aged 12 years old and above who own mobile phones and no mental or physical disabilities.
* Subjects willing to comply with given oral hygiene instructions.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-12-13 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Change in plaque index | At baseline and after 4 weeks.
  Plaque index: 0, no plaque, 1, plaque seen on the tip of the explorer or with disclosing agent, 2. plaque seen with the naked eye, 3, abundance of plaque.
Change in gingival index | At baseline and after 4 weeks.
  Gingival index: 0, normal gingiva, 1, mild inflammation - slight change in color, slight edema and no bleeding on probing, 2, moderate inflammation - redness, edema and glazing and bleeding on probing, 3, severe inflammation - marked redness and edema, ulceration and tendency to spontaneous bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Omar AlKadhi, BDS, MS, Principal Investigator — Riyadh Colleges of Dentistry and Pharmacy
Locations (1):
- Riyadh Colleges of Dentistry and Pharmacy, Riyadh, ArRiyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No